CLINICAL TRIAL: NCT04077437
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Site Phase 3 Study of the Efficacy and Safety of Manualized MDMA-Assisted Psychotherapy for the Treatment of Posttraumatic Stress Disorder of Moderate or Greater Severity
Brief Title: A Multi-Site Phase 3 Study of MDMA-Assisted Psychotherapy for PTSD (MAPP2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAPP2
Record Dates: First submitted 2019-08-30; First posted 2019-09-04 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Therapeutics; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind between group comparison of change in PTSD symptoms
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Use of separate databases for outcome measures and safety data. Assessment made by pool of independent raters. Randomization will be managed via an Interactive Web Randomization System (IWRS) based on a centralized randomization schedule developed by an independent thirdparty vendor to maintain blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: MDMA-assisted psychotherapy (Experimental): Administration of 80 to 120 mg midomafetamine HCl in combination with manualized psychotherapy, followed by a supplemental half-dose 1.5 to 2 hrs after the initial dose of 40 or 60 mg, respectively.
  Interventions: Behavioral: Therapy; Drug: Midomafetamine
- Placebo Comparator: Placebo (Placebo Comparator): Administration of inactive placebo in combination with manualized psychotherapy.
  Interventions: Behavioral: Therapy; Drug: Placebo

INTERVENTIONS:
Behavioral: Therapy — Standardized non-directive therapy performed by therapist team.
  Other Names: Manualized MDMA-assisted therapy
Drug: Midomafetamine — Administration of 80 to 120 mg midomafetamine HCl, followed by a supplemental half-dose 1.5 to 2 hrs after the initial dose of 40 or 60 mg, respectively, during three sessions of MDMA-assisted psychotherapy.
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA
  Arms: Experimental: MDMA-assisted psychotherapy
Drug: Placebo — Administration of placebo with therapy during three experimental sessions
  Other Names: Inactive placebo
  Arms: Placebo Comparator: Placebo

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective in people with at least moderate PTSD.

The main question it aims to answer is: Do three sessions of MDMA-assisted therapy reduce PTSD symptoms?

Researchers will compare three sessions of MDMA-assisted therapy with an initial dose of 80 to 120 mg to three sessions of placebo with therapy.

Participants will undergo three preparatory sessions without any study drug, followed by three MDMA-assisted therapy or placebo with therapy sessions. Each medication session will be followed by three integrative therapy sessions without study drug.

DETAILED DESCRIPTION:
This multi-site, double-blind, placebo-controlled, randomized Phase 3 study will assess the efficacy and safety of MDMA-assisted psychotherapy versus psychotherapy with placebo control in participants diagnosed with at least moderate PTSD. The study will be conducted in N ≈ 100 participants. Participants will be randomized into one of two groups (MDMA or placebo) in a 1:1 ratio. An initial dose of MDMA or placebo, followed by a supplemental half-dose unless contraindicated, will be administered during the Treatment Period with manualized psychotherapy in three monthly Experimental Sessions. This ~12-week Treatment Period is preceded by three Preparatory Sessions. Initial doses per Experimental Session include 80 mg or 120 mg of midomafetamine HCl or placebo followed 1.5 to 2 hours later by a supplemental half-dose (40 or 60 mg). Total amounts of midomafetamine HCl to be administered per Experimental Session range from 80 mg to 180 mg. Each Experimental Session will be followed by three Integrative Sessions of non-drug psychotherapy to help the participants process and understand their experiences during the Experimental Sessions.

The primary objective of this study is to evaluate the efficacy of MDMA-assisted psychotherapy for PTSD compared to identical psychotherapy with inactive placebo, as measured by change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Severity Score from Visit 3 (Baseline) to Visit 19 (18 weeks post Baseline) (Blake et al., 1995). The key secondary objective of this study is to evaluate the efficacy of MDMA-assisted psychotherapy for PTSD compared to identical psychotherapy with inactive placebo in clinician-rated functional impairment, as measured by the change in Sheehan Disability Scale (adapted SDS) item scores from Visit 3 (Baseline) to Visit 19 (18 weeks post Baseline) (Leon et al., 1997).

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Are fluent in speaking and reading the predominantly used or recognized language of the study site
* Are able to swallow pills
* Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments, and non-drug psychotherapy sessions
* Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session
* Must not participate in any other interventional clinical trials during the duration of the study
* Must be willing to remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures
* At baseline, have moderate PTSD diagnosis

Exclusion Criteria:

* Are not able to give adequate informed consent
* Have uncontrolled hypertension
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] in males and >460 ms in females corrected by Bazett's formula)
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Have evidence or history of significant medical disorders, such as myocardial infarction, cerebrovascular accident, or aneurysm
* Have symptomatic liver disease
* Have history of hyponatremia or hyperthermia
* Weigh less than 48 kilograms (kg)
* Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control
* Have an active illicit or prescription drug use disorder
* Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session; or have previously participated in a MAPS-sponsored MDMA clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (12):
  - New School Research, Los Angeles, California
  - San Francisco Insight and Integration Center, San Francisco, California
  - UCSF, San Francisco, California
  - Aguazul Bluewater, Inc., Boulder, Colorado
  - Wholeness Center, Fort Collins, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Ray Worthy Psychiatry LLC, New Orleans, Louisiana
  - Trauma Research Foundation, Boston, Massachusetts
  - New York University, New York, New York
  - Nautilus Psychiatric Services, New York, New York
  - Zen Therapeutic Solutions, LLC, Mt. Pleasant, South Carolina
  - University of Wisconsin - Madison, Madison, Wisconsin
- Israel (2):
  - Assaf Harofeh Research Fund, Beer Yaaqov
  - Sheba Fund for Health Services and Research, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when the database has been locked and data has been unblinded.
Access Criteria: Interested persons should correspond with the central contact for the multisite study.

REFERENCES:
- [Background] Leon AC, Olfson M, Portera L, Farber L, Sheehan DV. Assessing psychiatric impairment in primary care with the Sheehan Disability Scale. Int J Psychiatry Med. 1997;27(2):93-105. doi: 10.2190/T8EM-C8YH-373N-1UWD. PMID 9565717
- [Background] Blake DD, Weathers FW, Nagy LM, Kaloupek DG, Gusman FD, Charney DS, Keane TM. The development of a Clinician-Administered PTSD Scale. J Trauma Stress. 1995 Jan;8(1):75-90. doi: 10.1007/BF02105408. PMID 7712061
- [Derived] Mitchell JM, Ot'alora G M, van der Kolk B, Shannon S, Bogenschutz M, Gelfand Y, Paleos C, Nicholas CR, Quevedo S, Balliett B, Hamilton S, Mithoefer M, Kleiman S, Parker-Guilbert K, Tzarfaty K, Harrison C, de Boer A, Doblin R, Yazar-Klosinski B; MAPP2 Study Collaborator Group. MDMA-assisted therapy for moderate to severe PTSD: a randomized, placebo-controlled phase 3 trial. Nat Med. 2023 Oct;29(10):2473-2480. doi: 10.1038/s41591-023-02565-4. Epub 2023 Sep 14. PMID 37709999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through print and internet advertisements, referrals from other treatment providers, and by word of mouth.
Groups:
- Experimental: MDMA-assisted Psychotherapy: Administration of 80 to 120 mg midomafetamine HCl in combination with psychotherapy, followed by a supplemental half-dose of 40 or 60 mg offered 1.5 to 2 hrs after the initial dose, respectively.
- Placebo Comparator: Placebo With Psychotherapy: Administration of inactive placebo in combination with psychotherapy.
Period: Overall Study
Arm/Group | Experimental: MDMA-assisted Psychotherapy | Placebo Comparator: Placebo With Psychotherapy
Started | 53 | 51
Completed | 52 | 42
Not Completed | 1 | 9

BASELINE CHARACTERISTICS:
Groups:
- Experimental: MDMA-assisted Psychotherapy: Administration of 80 to 120 mg MDMA in combination with psychotherapy, followed by a supplemental half-dose of 40 or 60 mg MDMA offered 1.5 to 2 hrs after the initial dose, respectively.
  Behavioral: Psychotherapy: Standardized non-directive psychotherapy performed by therapist team.
  MDMA: Administration of 80 to 120 mg MDMA during three sessions of MDMA-assisted psychotherapy, followed by a supplemental half-dose of 40 or 60 mg MDMA offered 1.5 to 2 hrs after the initial dose, respectively.
- Placebo Comparator: Placebo With Psychotherapy: Administration of inactive placebo in combination with psychotherapy.
  Behavioral: Psychotherapy: Standardized non-directive psychotherapy performed by therapist team.
  Placebo: Administration of placebo during three sessions of MDMA-assisted psychotherapy.
- Total: Total of all reporting groups
Arm/Group | Experimental: MDMA-assisted Psychotherapy | Placebo Comparator: Placebo With Psychotherapy | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (11.0) | 39.9 (9.6) | 39.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 42 | 74
  Male | 21 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 11 | 28
  Not Hispanic or Latino | 36 | 39 | 75
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  White | 37 | 32 | 69
  More than one race | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Baseline PTSD Duration [Mean (Standard Deviation); unit: years] | 16.3 (14.3) | 16.1 (12.4) | 16.2 (13.3)
Baseline CAPS-5 Dissociative Subtype [Count of Participants; unit: Participants] | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Primary Endpoint in Clinician Administered PTSD Scale for DSM-V (CAPS-5)
Description: The CAPS-5 is a 30-item semi-structured interview assessing PTSD in the past month through diagnostic and symptom severity scores anchored to a DSM-5 defined traumatic event. The CAPS-5 produces a Total Severity Score based on severity of PTSD domains described in the DSM-5, as well as a categorical rating indicating whether a participant meets PTSD diagnostic criteria. CAPS-5 Total Symptom Severity scores range from 0 to 80 with higher values indicating greater symptom severity. CAPS-5 assigns PTSD diagnosis as being present or absent.
Time Frame: Baseline to 18 weeks post baseline post enrollment confirmation
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Experimental: MDMA-assisted Psychotherapy | Placebo Comparator: Placebo With Psychotherapy
Number analyzed (Participants) | 53 | 50
score on a scale | -23.69 [-26.94 to -20.44] | -14.78 [-18.28 to -11.28]

2. Secondary Outcome: Change From Baseline to Primary Endpoint in Adapted Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a clinician-rated assessment of functional impairment that was adapted for the purposes of this study to limit missing item-level data as per the FDA requirements and included use of the three-item mean as the total score and imputation of work-related impairment. The SDS is a 3-item scale measuring the severity of disability in the domains of work, family life/home responsibilities and social/leisure activities, with each item scored on a ten-point Likert scale from 0 ('not at all impaired') to 10 ('very severely impaired'). The SDS total score was the mean of the 3 item responses. The SDS total score ranged from 0 to 10, with higher scores indicating greater functional impairment.
Time Frame: Baseline to 18 weeks post enrollment confirmation
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Placebo Comparator: Placebo: Administration of inactive placebo in combination with psychotherapy.
  Behavioral: Psychotherapy: Standardized non-directive psychotherapy performed by therapist team.
  Placebo: Administration of placebo during three sessions of MDMA-assisted psychotherapy.
Arm/Group | Experimental: MDMA-assisted Psychotherapy | Placebo Comparator: Placebo
Number analyzed (Participants) | 53 | 50
score on a scale | -3.31 [-4.03 to -2.60] | -2.11 [-2.89 to -1.33]

ADVERSE EVENTS:
Time Frame: During the Treatment Period from the first Experimental Session to the last Integrative Session (approximately 12 weeks)
Groups:
- MDMA-assisted Therapy: Administration of 80 to 120 mg midomafetamine HCl in combination with psychotherapy, followed by a supplemental half-dose of 40 or 60 mg offered 1.5 to 2 hrs after the initial dose, respectively.
- Placebo With Therapy: Administration of inactive placebo in combination with psychotherapy.
Arm/Group | MDMA-assisted Therapy | Placebo With Therapy
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/51
Other Adverse Events (participants affected / at risk) | 53/53 | 49/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MDMA-assisted Therapy (N=53) | Placebo With Therapy (N=51)
Palpitations (Cardiac disorders) | 5 | 1
Vision blurred (Eye disorders) | 8 | 0
Mydriasis (Eye disorders) | 6 | 0
Visual impairment (Eye disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 24 | 11
Dry mouth (Gastrointestinal disorders) | 9 | 4
Abdominal discomfort (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 14 | 9
Feeling hot (General disorders) | 14 | 6
Feeling cold (General disorders) | 11 | 3
Chest discomfort (General disorders) | 9 | 2
Chills (General disorders) | 8 | 1
Feeling jittery (General disorders) | 8 | 0
Feeling abnormal (General disorders) | 5 | 2
Feeling of body temperature change (General disorders) | 5 | 0
Thirst (General disorders) | 4 | 1
Gait disturbance (General disorders) | 3 | 0
COVID-19 (Infections and infestations) | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Heart rate increased (Investigations) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 19 | 5
Muscle tightness (Musculoskeletal and connective tissue disorders) | 31 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Pain in jaw (Musculoskeletal and connective tissue disorders) | 6 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0
Headache (Nervous system disorders) | 38 | 31
Dizziness (Nervous system disorders) | 15 | 8
Paraesthesia (Nervous system disorders) | 10 | 1
Nystagmus (Nervous system disorders) | 7 | 1
Disturbance in attention (Nervous system disorders) | 3 | 3
Hypoaesthesia (Nervous system disorders) | 5 | 1
Tremor (Nervous system disorders) | 6 | 0
Suicidal ideation (Psychiatric disorders) | 18 | 21
Insomnia (Psychiatric disorders) | 19 | 15
Anxiety (Psychiatric disorders) | 15 | 12
Depressed mood (Psychiatric disorders) | 5 | 6
Restlesness (Psychiatric disorders) | 8 | 2
Bruxism (Psychiatric disorders) | 7 | 1
Nightmare (Psychiatric disorders) | 4 | 3
Emotional disorder (Psychiatric disorders) | 3 | 2
Irritability (Psychiatric disorders) | 3 | 2
Panic attack (Psychiatric disorders) | 3 | 1
Binge eating (Psychiatric disorders) | 0 | 3
Dissociation (Psychiatric disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 18 | 3
Flushing (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04077437/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT04077437/SAP_001.pdf
  • Informed Consent Form (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04077437/ICF_003.pdf